CLINICAL TRIAL: NCT05697510
Title: Monocentric Phase 1 Study With Dose-escalation of Siltuximab in Combination With Idarubicin and Cytarabine Chemotherapy in Patients With Acute Myeloblastic Leukaemia (AML) With Poor Prognosis: SILTUXILAM
Brief Title: Dose-escalation of Siltuximab in Combination With Idarubicin and Cytarabine Chemotherapy in Patients With Acute Myeloblastic Leukaemia (AML) With Poor Prognosis: SILTUXILAM
Acronym: SILTUXILAM
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RC22_0233; 2022-501171-14-00 (Other: EU CT number)
Record Dates: First submitted 2023-01-11; First posted 2023-01-26 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: AML IL-6 SILTUXIMAB
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — siltuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SILTUXIMAB (Experimental)
  Interventions: Drug: Siltuximab

INTERVENTIONS:
Drug: Siltuximab — Administration of siltuximab at day 8 of induction following a classical induction; 3 dose levels : 7, 9 and 11mg/kg

SUMMARY:
This is a phase 1 dose escalation study testing the addition of an anti-IL6 (siltuximab) to standard induction chemotherapy for high-risk AML.

DETAILED DESCRIPTION:
Administration of siltuximab at day 8 of induction following a classical induction using idarubicin 8mg/m2/d for 5 days and cytarabine 100mg/m2/d for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* age >= 18 years
* AML with a poor prognosis defined according to the criteria below:

LAM First line: Age <60 years and unfavorable risk according to the 2017 ELN Age> = 60 years old and intermediate or unfavorable risk according to the ELN 2017 LAM in Relapse: whatever the age

* ECOG <= 2
* Patient eligible for intensive chemotherapy
* Informed consent
* Liver function tests: transaminases <3x normal, bilirubin <1.5X normal
* Creatinine clearance> 60ml / min
* LVEF> = 50%

Exclusion Criteria:

* Patients with FLT3 ITD or TKD mutation eligible for FLT3 inhibitor therapy
* Uncontrolled infection
* Hep B, C, HIV +
* History of diverticulosis / diverticulitis
* Patients at high risk of gastrointestinal perforation
* No social security or any other scheme
* Pregnant women or patient unable to take contraception (pill, abstinence, IUD not allowed) in case of fertility. contraceptive pill, abstinence, unauthorised IUD) in case of fertility. A patient who cannot continue contraception for at least 3 months after the last SILTUXIMAB injection is not eligible for inclusion.
* Lactating women
* Minors
* Adults under guardianship, curatorship or legal protection
* Hypersensitivity to one of the active substances or to one of the excipients

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-03-16 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
number of DLT | 45 days

SECONDARY OUTCOMES:
Evaluation of the response to induction therapy with idarubicin + cytarabine + siltuximab | Day 30 and Day 45
  Calculation of complete remission (CR) and CR with incomplete recovery (CRi) according to the ELN 2017 definition
Evaluation of response at D15 after induction | Day 15
  percent bone marrow blasts at D15 (myelogram)
Assessment of myelotoxicity | Day 45
  Neutrophil recovery time (>1.0 × 109/L) from D1; Platelet recovery time (>100 × 109/L) from D1
Overall survival | Month 6
  delay from D1 of induction to date of last news or death
Leukaemia-free survival | Month 6
  delay between the date of CR and the date of relapse or death or the date of the last follow-up
Event-free survival | Month 6
  delay between D1 of induction and the date of relapse, death or date of last
Incidence of relapse if remission | Month 6
  relapse rate at last follow-up
Infections | Month 6
  monitoring of AEs infection
Cytokine levels: FLT3L and IL-6 | Day 1, Day 8, Day 15, Day 22
  Cytokine levels: FLT3L and IL-6

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: No